CLINICAL TRIAL: NCT06405269
Title: A Multicentre Prospective Cohort Study: Effect of (neo)Adjuvant Therapy on Lipids in Young Breast Cancer Patients
Brief Title: Effect of (neo)Adjuvant Therapy on Lipids in Young Breast Cancer Patients
Status: Enrolling by invitation | Type: Observational
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, PENG YUAN, Professor, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Other Study IDs: NCC3872
Record Dates: First submitted 2024-05-04; First posted 2024-05-08 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2024-05

CONDITIONS: Breast Neoplasms; Lipid Profile
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Regular blood tests are performed to monitor the patient's lipid profile
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Adjuvant chemotherapy group（Hormone receptor negative breast cancer）: Patients receiving adjuvant chemotherapy after surgery for hormone receptor-negative breast cancer
- Adjuvant chemotherapy group（Hormone receptor positive breast cancer）: Patients receiving adjuvant chemotherapy after surgery for hormone receptor-positive breast cancer
- Without adjuvant chemotherapy group（Hormone receptor positive breast cancer）: Patients without adjuvant chemotherapy after surgery for hormone receptor-positive breast cancer

SUMMARY:
Previous studies have shown differences in the effects of different endocrine drugs on blood lipids in breast cancer, and dyslipidaemia is a major risk factor for cardiovascular disease, and it has been previously reported that the leading cause of death in postmenopausal patients with breast cancer is cardiovascular disease, but the effects of endocrine drug therapy on blood lipids in young breast cancer patients (age ≤40) are not clear. Previously, our group conducted a preliminary retrospective analysis of young patients on endocrine therapy and found that dyslipidaemia was also a common adverse effect of treatment in young breast cancer patients; therefore, dyslipidaemia induced by antineoplastic therapy not only occurs in postmenopausal patients, but is also prevalent in premenopausal and even younger patients. Therefore, this study intends to evaluate the effects of different treatment regimens on lipids in early-stage young breast cancer patients and to explore the optimal timing of lipid-lowering drug interventions to provide a basis for clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* ECOG score 0-1
* Resectable breast cancer
* No distant metastases on postoperative imaging assessment
* Patients proposed for (neo)adjuvant therapy
* No previous oral lipid-lowering drugs, serum LDL-C level within normal range, i.e. LDL-C value: <3.4 mmol/L
* No fatty liver by liver ultrasound/CT examination
* No major organ dysfunction

Exclusion Criteria:

* Patients with pre-existing hyperlipidaemia, coronary heart disease, fatty liver disease, or who have received or are receiving lipid-lowering medication
* Enrolled in another study or less than or equal to 4 weeks since discontinuation of other medications
* Presence of severe dysfunction of vital organs
* Patients with other malignancies (except cured non-melanoma skin cancer, cervical carcinoma in situ and other tumours that have been cured for at least 5 years)
* Acute infectious diseases or chronic infectious diseases in active stage
* History of uncontrolled epilepsy, central nervous system disease or mental disorder

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Young breast cancer patients who fulfil the following criteria: less than or equal to 40, surgically resectable, requiring (neo)adjuvant chemotherapy or endocrine therapy.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2024-05-06 (Actual); Primary Completion 2029-05-01 (Estimated); Study Completion 2029-05-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who developed LDL-C abnormalities in 3 groups | 2 years
  Observe and compare differences between groups

SECONDARY OUTCOMES:
Proportion of patients who developed TC，LDL-C，and TG abnormalities in 3 groups | 2 years
  Observe and compare differences between groups
Proportion of patients developing fatty liver in 3 groups | 2 years
  Observe and compare differences between groups

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No